CLINICAL TRIAL: NCT00235313
Title: Does Dose Adjustment of Nicotine Replacement Therapies According to Saliva Cotinine Increase Efficacy of These Treatments of Assistance To the Nicotinic Weaning Of the High-Risk Patients?
Brief Title: Adjustment of DOses of NIcotine in Smoking Cessation (ADONIS)
Acronym: ADONIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Health Products Safety Agency (Other Government)
Responsible Party: Christophe AUCAN, Department of Clinical Trial of Developpement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P040406; AOR04001
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2007-03

CONDITIONS: Smoking Cessation
Keywords: Nicotine replacement therapies; Smoking; Smoking related diseases; Saliva cotinine; Dose adjustment; Smoker; patients with smoking related disease conditions
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): adaptation of the nicotine patch with salivary cotinine
  Interventions: Procedure: Dose adjustment of nicotine replacement therapies
- 2 (Other): normal following with a nicotine patch
  Interventions: Drug: nicotine patch

INTERVENTIONS:
Procedure: Dose adjustment of nicotine replacement therapies — Dose adjustment of nicotine replacement therapies
  Arms: 1
Drug: nicotine patch — normal following with a nicotine patch
  Other Names: normal following with a nicotine patch
  Arms: 2

SUMMARY:
Nicotine replacement therapies (NRT) have proven efficacy to help smokers quit. However, their effectiveness is low. This study aims to answer the question: Does the dose adjustment of NRT according the saliva concentration of nicotine's main metabolite: cotinine improve their efficacy compared with the lack of dose adjustment (usual care) in smoking patients with smoking related disease condition.

DETAILED DESCRIPTION:
Smokers currently smoking at least 10 cigarettes per day with smoking related diseases are included. They are randomized either to receive standard nicotine replacement therapy (24 h nicotine patch 21, 14, 7 mg/day for one month each, respectively), control arm, or nicotine dose adjustment according their saliva cotinine: dose adaptation arm. In the control arm, at the discretion of the investigators, buccal forms of nicotine replacement therapies are allowed. In both arms, saliva cotinine determinations are performed every 2 weeks for 2 months. In the control arm saliva cotinine results are not communicated to the investigators. In the dose adaptation arm investigators receive saliva cotinine results and should adapt the nicotine doses (mg of nicotine/day) according to baseline (when smoking) saliva cotinine to obtain 100 % substitution. Smokers are assessed at weekly visits after the predetermined quit day for 3 months. Follow up at 6 months. Main outcome measure: sustained abstinence (self reported no smoking and expired air carbon monoxide concentration equal or less than 8 ppm during the last (3rd) month of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years Smoking ≥ 10 cigarettes per day Patients with disease conditions known to be related to smoking: e.g.coronary heart diseases, COPD, lower extremity arterial disease, etc

Exclusion Criteria:

* Smokers whose follow-up during the duration of the study, in a predictable way, cannot be assured.
* smokers having been treated by bupropion ( Zyban) during two months preceding the inclusion
* persons under TSN, neuroleptic, substitute treatments in OPINOIDES, under anticoagulants-non-equilibrating,
* encircled woman
* breast-feeding woman
* Contraindication usual of the TSN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
sustained smoking abstinence | during the study

SECONDARY OUTCOMES:
point prevalence abstinence,craving for tobacco,symptoms of nicotine withdrawal,weight,saliva cotinine concentration,genetic polymorphisms as predictors of therapeutic response and in interaction with nicotine replacement therapies | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Yvan BERLIN, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Unité de Recherche Clinique, Paris, France

REFERENCES:
- [Background] Dale LC, Hurt RD, Offord KP, Lawson GM, Croghan IT, Schroeder DR. High-dose nicotine patch therapy. Percentage of replacement and smoking cessation. JAMA. 1995 Nov 1;274(17):1353-8. PMID 7563559
- [Derived] Berlin I, Singleton EG, Heishman SJ. Cross validation of the prognostic and diagnostic utility of tobacco craving in a general and a pregnant sample of treatment-seeking smokers. Drug Alcohol Depend. 2015 Sep 1;154:174-83. doi: 10.1016/j.drugalcdep.2015.06.034. Epub 2015 Jun 29. PMID 26160457
- [Derived] Berlin I, Singleton EG, Heishman SJ. Predicting smoking relapse with a multidimensional versus a single-item tobacco craving measure. Drug Alcohol Depend. 2013 Oct 1;132(3):513-20. doi: 10.1016/j.drugalcdep.2013.03.017. Epub 2013 Apr 23. PMID 23623506
- [Derived] Berlin I, Jacob N, Coudert M, Perriot J, Schultz L, Rodon N. Adjustment of nicotine replacement therapies according to saliva cotinine concentration: the ADONIS* trial-a randomized study in smokers with medical comorbidities. Addiction. 2011 Apr;106(4):833-43. doi: 10.1111/j.1360-0443.2010.03306.x. Epub 2011 Feb 14. PMID 21205047